CLINICAL TRIAL: NCT05826574
Title: A Phase 1, Open Label, Fixed Sequence Study to Assess the Pharmacokinetics of Brensocatib When Administered Alone and With Multiple Doses of Rifampin (CYP3A Inducer) or Esomeprazole (Proton Pump Inhibitor) in Healthy Subjects
Brief Title: A Study to Assess Pharmacokinetics (PK) of Brensocatib Alone and With Multiple Doses of Rifampin or Esomeprozole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS1007-106
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
Keywords: Brensocatib; INS1007
MeSH Terms: interventions — brensocatib; Rifampin; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Period 1: Brensocatib (Experimental): Period 1: Participants will receive a single oral dose of brensocatib on Day 1 in Part 1 of the study.
  Interventions: Drug: Brensocatib
- Part 1: Period 2: Brensocatib + Rifampin (Experimental): Period 2: Participants will receive rifampin 600 mg once daily (QD), orally, on Days 8 to 23 along with a single oral dose of brensocatib prior to the rifampin administration on Day 17 in Part 1 of the study.
  Interventions: Drug: Brensocatib; Drug: Rifampin
- Part 2: Period 1: Brensocatib (Experimental): Period 1: Participants will receive a single oral dose of brensocatib on Day 1 in Part 2 of the study.
  Interventions: Drug: Brensocatib
- Part 2: Period 2: Brensocatib + Esomeprazole (Experimental): Period 2: Participants will receive esomeprazole 40 mg QD, orally, on Days 8 to 12 along with a single oral dose of brensocatib prior to the esomeprazole administration on Day 12 in Part 2 of the study.
  Interventions: Drug: Brensocatib; Drug: Esomeprazole

INTERVENTIONS:
Drug: Brensocatib — Oral tablets.
  Other Names: INS1007
Drug: Rifampin — Oral capsules.
  Arms: Part 1: Period 2: Brensocatib + Rifampin
Drug: Esomeprazole — Oral capsules.
  Arms: Part 2: Period 2: Brensocatib + Esomeprazole

SUMMARY:
The primary purpose of this study is to assess the effects of rifampin on the PK of brensocatib in Part 1 of the study and to assess the effects of esomeprazole on the PK of brensocatib in Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants defined by no significant other conditions as in the protocol.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, immunological, oncologic, or psychiatric disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, as determined by the investigator (or designee).

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-07-16 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 2: Area Under the Concentration-time (AUC) of Brensocatib in Plasma | Pre-dose and at multiple timepoints post-dose on Days 1 to 7, 17 (Part 1), and Days 1 to 7, 12 to 18 (Part 2)
  Pharmacokinetics of brensocatib following a single dose in healthy participants will be assessed.

SECONDARY OUTCOMES:
Parts 1 and 2: Number of Participants Who Experienced at Least One Adverse Event (AE) | Up to Day 31 (Part 1) and up to Day 26 (Part 2)
  Safety and tolerability of brensocatib when administered alone and in combination with rifampin/esomeprazole will be determined in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No